CLINICAL TRIAL: NCT00163969
Title: The Use of Ketamine as Rescue Analgesia in the Recovery Room Following Opioid Administration. A Double-blind Randomised Trial in Postoperative Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161/01
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2005-09

CONDITIONS: Post Operative Pain
Keywords: Pain; Wind-up; opioid; ketamine; pre-emptive
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
This clinical trial will determine if postoperative patients who have postoperative pain, which has been refractory to morphine administration, will have improved pain relief following a bolus administration of ketamine as compared with an ongoing morphine dosing regimen

DETAILED DESCRIPTION:
Some patients require large doses of opioids to control postoperative pain, which can result in a prolonged period of poor pain control, and potentially increased side effects associated with large morphine doses. This may be due to insufficient morphine dose to that individual or acute tolerance ( 1 ). Ketamine is not just an anaesthetic agent but at lower doses is known to provide efficacious analgesia ( 2, 3 ). Ketamine has been shown to have a marked analgesic effect on high intensity nociceptive stimuli ( 4 ) as exhibited in postoperative pain. When given for opioid analgesia resistant cancer pain in bolus doses at two different concentrations it has been shown to be effective and have a morphine-sparing effect, without undue complications ( 5 ).

Ketamine has been suggested to work pre-emptively and also by many other routes other than intravenously ( 6 - 9 ) .

Previous studies have compared morphine with morphine and ketamine administered as PCA or intramuscularly ( 10 - 12 ) in postoperative patients with varying effects. Javery et al. ( 11 ) showed that pain scores were lower in patients who received ketamine but Reeves et al. in a later but similar study showed no significant difference ( 13 ).

The authors have noted that in the postoperative situation with morphine resistant pain, a bolus dose of ketamine not only leads to a marked decline in pain but it also remains efficacious for several hours. This prolonged effect was also noted in opioid resistant cancer pain ( 5 ). This indeed may have relevance to the prevention of onset of chronic post surgical pain ( 14 ) and earlier discharge from the Post Anaesthetic Care Unit.

Morphine and ketamine are not without side effects. Respiratory depression, nausea, vomiting and vivid dreams, being well documented will hence be a secondary endpoint. A quality of recovery score will also be measured ( 15 ) and four hours postoperatively.

This study is designed to compare a morphine regimen in the form of a standard Post Anaesthetic Care Unit pain protocol with a bolus dose of ketamine to be implemented if the pain protocol has been inadequate. Any patient in pain, despite two doses of morphine will be included. Thereafter the patients will be randomised to receive either a further solution of ketamine or continuation of the morphine protocol. This randomised, double-blinded, trial will be based in the Post Anaesthetic Care Unit under close anaesthetic and nursing staff supervision.

ELIGIBILITY:
Inclusion Criteria:

* 1. Those patients requiring the routine pain protocol to be implemented as used in the Post Anaesthetic Care Unit who need more than two doses of morphine (and having received intraoperative morphine).

Exclusion Criteria:

* Exclusion Criteria

  1. Known allergy to morphine or ketamine.
  2. Past history of major psychiatric disturbance or currently taking psychiatric medication/s.
  3. Chronic morphine usage.
  4. Chronic pain syndrome or chronic painful medical condition.
  5. Unable to obtain a reliable pain score in recovery due to language barriers or residual anaesthesia.
  6. Known pregnancy.
  7. Cases where primary anaesthetist prefers alternate therapy.
  8. Aged less than 18 years.
  9. Weight less than 50 kilograms or greater than 100 kilograms.
  10. Use of ketamine intraoperatively.
  11. Use of major regional block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04; Study Completion 2004-09

PRIMARY OUTCOMES:
Pain scores at rest in recovery and at four hours postoperatively

SECONDARY OUTCOMES:
Morphine protocol consumption.
Sedation scores - Recovery Room and four hours.
PONV scores - Recovery Room and four hours.
Frequency of antiemetic administration - Recovery Room and up to four hours.
Quality of recovery score preoperatively and at four hours.
Adverse events (vivid dreams, nausea, hallucinations, respiratory depression, pruritus) - Recovery Room and at four hours.
Time to discharge from the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: David E Lindholm, MBBS FANZCA, Principal Investigator — The Alfred
Locations (1):
- The Alfred Commercial Rd Prahran, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Mercadante S, Portenoy RK. Opioid poorly-responsive cancer pain. Part 2: basic mechanisms that could shift dose response for analgesia. J Pain Symptom Manage. 2001 Mar;21(3):255-64. doi: 10.1016/s0885-3924(00)00236-0. PMID 11239748
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Macrae W A, Davies H T O Chronic post surgical pain Epidemiology of Pain edited by Crombie I K. IASP Press. Seattle 1999. 125 - 142
- [Background] Reeves M, Lindholm DE, Myles PS, Fletcher H, Hunt JO. Adding ketamine to morphine for patient-controlled analgesia after major abdominal surgery: a double-blinded, randomized controlled trial. Anesth Analg. 2001 Jul;93(1):116-20. doi: 10.1097/00000539-200107000-00025. PMID 11429351
- [Background] Marcus RJ, Victoria BA, Rushman SC, Thompson JP. Comparison of ketamine and morphine for analgesia after tonsillectomy in children. Br J Anaesth. 2000 Jun;84(6):739-42. doi: 10.1093/oxfordjournals.bja.a013585. PMID 10895748
- [Background] Javery KB, Ussery TW, Steger HG, Colclough GW. Comparison of morphine and morphine with ketamine for postoperative analgesia. Can J Anaesth. 1996 Mar;43(3):212-5. doi: 10.1007/BF03011736. PMID 8829857
- [Background] Adriaenssens G, Vermeyen KM, Hoffmann VL, Mertens E, Adriaensen HF. Postoperative analgesia with i.v. patient-controlled morphine: effect of adding ketamine. Br J Anaesth. 1999 Sep;83(3):393-6. doi: 10.1093/bja/83.3.393. PMID 10655908
- [Background] Schmid RL, Sandler AN, Katz J. Use and efficacy of low-dose ketamine in the management of acute postoperative pain: a review of current techniques and outcomes. Pain. 1999 Aug;82(2):111-125. doi: 10.1016/S0304-3959(99)00044-5. PMID 10467917
- [Background] Azevedo VM, Lauretti GR, Pereira NL, Reis MP. Transdermal ketamine as an adjuvant for postoperative analgesia after abdominal gynecological surgery using lidocaine epidural blockade. Anesth Analg. 2000 Dec;91(6):1479-82. doi: 10.1097/00000539-200012000-00034. PMID 11094004
- [Background] Aida S, Yamakura T, Baba H, Taga K, Fukuda S, Shimoji K. Preemptive analgesia by intravenous low-dose ketamine and epidural morphine in gastrectomy: a randomized double-blind study. Anesthesiology. 2000 Jun;92(6):1624-30. doi: 10.1097/00000542-200006000-00020. PMID 10839912
- [Background] Stubhaug A, Breivik H, Eide PK, Kreunen M, Foss A. Mapping of punctuate hyperalgesia around a surgical incision demonstrates that ketamine is a powerful suppressor of central sensitization to pain following surgery. Acta Anaesthesiol Scand. 1997 Oct;41(9):1124-32. doi: 10.1111/j.1399-6576.1997.tb04854.x. PMID 9366932
- [Background] Mercadante S, Arcuri E, Tirelli W, Casuccio A. Analgesic effect of intravenous ketamine in cancer patients on morphine therapy: a randomized, controlled, double-blind, crossover, double-dose study. J Pain Symptom Manage. 2000 Oct;20(4):246-52. doi: 10.1016/s0885-3924(00)00194-9. PMID 11027905
- [Background] Arendt-Nielsen L, Petersen-Felix S, Fischer M, Bak P, Bjerring P, Zbinden AM. The effect of N-methyl-D-aspartate antagonist (ketamine) on single and repeated nociceptive stimuli: a placebo-controlled experimental human study. Anesth Analg. 1995 Jul;81(1):63-8. doi: 10.1097/00000539-199507000-00013. PMID 7598284
- [Background] Owen H, Reekie RM, Clements JA, Watson R, Nimmo WS. Analgesia from morphine and ketamine. A comparison of infusions of morphine and ketamine for postoperative analgesia. Anaesthesia. 1987 Oct;42(10):1051-6. doi: 10.1111/j.1365-2044.1987.tb05167.x. PMID 3318543
- [Background] Clements JA, Nimmo WS. Pharmacokinetics and analgesic effect of ketamine in man. Br J Anaesth. 1981 Jan;53(1):27-30. doi: 10.1093/bja/53.1.27. PMID 7459184